CLINICAL TRIAL: NCT05632263
Title: Evaluate the Predictive Impact of the EHMRG Score for Patients Admitted to the Emergency Department With Final Diagnosis of Acute Heart Failure
Brief Title: Evaluate the Predictive Impact of the EHMRG
Acronym: EHMRGscore
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, clinical proffesor, University of Monastir
Other Study IDs: EHMRG_MIR
Record Dates: First submitted 2022-11-19; First posted 2022-11-30 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Emergencies; Heart Diseases
Keywords: EHMRGscore; ACUTE HEART FAILURE
MeSH Terms: conditions — Emergencies; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EHMRGscore: validation of the EHMRG score for hospitalized patients with acute heart failure in the emergency department
  Interventions: Diagnostic Test: EHMRGscore

INTERVENTIONS:
Diagnostic Test: EHMRGscore — validation of the EHMRG score for hospitalized patients with acute heart failure in the emergency department

SUMMARY:
External validation of the EHMRG score for hospitalized patients with acute heart failure in the emergency department

DETAILED DESCRIPTION:
It is a prospective cohort study carried out in the ED of Monastir which included patients admitted to the ED with a discharge diagnosis of AHF.

ELIGIBILITY:
Inclusion Criteria:

* Patients consulted for acute dyspnea and were diagnosed with acute heart failure.
* Major patient.
* Subject who accept to participate in the research.

Exclusion Criteria:

* Patient who refuse to participate in the study.
* Impossibility of giving the patient informed information

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is a prospective cohort study carried out in the ED of Monastir over a period from February 2009 to September 2020 which included patients admitted to the ED with a discharge diagnosis of AHF.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
EHMRGscore | 7days
  The primary outcome of interest is the EHMRG predictive accuracy to prognosticate 7-day mortality was measured by the athe area under the receiver operating characteristic curver (AUROC) with 95% confidence intervals.

SECONDARY OUTCOMES:
Re-admission rate 30-day re-admission rate | 30days
  30day ré-admission rate
Mortality rate Mortality rate at 30 days | 30day
  Mortality rate at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Pr, Principal Investigator — University of Monastir

IPD SHARING:
Plan to Share IPD: No
The EHMRG Risk score is based on commonly available parameters at presentation.
  It includes 10 predictors of mortality: age/mode of ED presentation / SBP / heart-rate / oxygen saturation/potassium concentration, creatinine concentration, troponin, presence of active cancer, and treatment with metolazone.